CLINICAL TRIAL: NCT00963157
Title: A Phase II Study in Healthy Adult and Elderly Populations to Assess the Safety and Immunogenicity of a Sanofi Pasteur H1N1 Influenza Vaccine Administered at Different Dose Levels Given With and Without GlaxoSmithKline AS03 Adjuvant
Brief Title: Sanofi H1N1 Influenza Vaccine Administered at Different Dose Levels With and Without AS03 Adjuvant in Healthy Adult and Elderly Populations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 09-0058
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Results first posted 2011-12-14 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2011-01

CONDITIONS: Influenza
Keywords: H1N1, influenza A viruses, vaccine, elderly
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (5):
- Group 1: 3.75 mcg H1N1 vaccine + AS03 adjuvant (Experimental): 150 subjects (100 aged 18-64 and 50 aged greater than or equal to 65) to receive 3.75 mcg H1N1 vaccine plus AS03 adjuvant on Day 0 and Day 21.
  Interventions: Drug: AS03; Biological: Influenza Virus Vaccine, Monovalent A/H1N1 A/California/7/2009 NYMC X-179A
- Group 5: 15 mcg H1N1 vaccine unadjuvanted (Experimental): 150 subjects (100 aged 18-64 and 50 aged greater than or equal to 65) to receive 15 mcg H1N1 vaccine unadjuvanted on Day 0 and Day 21.
  Interventions: Biological: Influenza Virus Vaccine, Monovalent A/H1N1 A/California/7/2009 NYMC X-179A
- Group 4: 7.5 mcg H1N1 vaccine unadjuvanted (Experimental): 150 subjects (100 aged 18-64 and 50 aged greater than or equal to 65) to receive 7.5 mcg H1N1 vaccine unadjuvanted on Day 0 and Day 21.
  Interventions: Biological: Influenza Virus Vaccine, Monovalent A/H1N1 A/California/7/2009 NYMC X-179A
- Group 2: 7.5 mcg H1N1 vaccine + AS03 adjuvant (Experimental): 150 subjects (100 aged 18-64 and 50 aged greater than or equal to 65) to receive 7.5 mcg H1N1 vaccine plus AS03 adjuvant on Day 0 and Day 21.
  Interventions: Drug: AS03; Biological: Influenza Virus Vaccine, Monovalent A/H1N1 A/California/7/2009 NYMC X-179A
- Group 3: 15 mcg H1N1 vaccine + AS03 adjuvant (Experimental): 150 subjects (100 aged 18-64 and 50 aged greater than or equal to 65) to receive 15 mcg H1N1 vaccine plus AS03 adjuvant on Day 0 and Day 21.
  Interventions: Drug: AS03; Biological: Influenza Virus Vaccine, Monovalent A/H1N1 A/California/7/2009 NYMC X-179A

INTERVENTIONS:
Drug: AS03 — AS03 adjuvant administered with 3.75, 7.5, or 15 mcg inactivated H1N1 vaccine.
  Arms: Group 1: 3.75 mcg H1N1 vaccine + AS03 adjuvant; Group 2: 7.5 mcg H1N1 vaccine + AS03 adjuvant; Group 3: 15 mcg H1N1 vaccine + AS03 adjuvant
Biological: Influenza Virus Vaccine, Monovalent A/H1N1 A/California/7/2009 NYMC X-179A — Inactivated influenza H1N1 vaccine with AS03 adjuvant, delivered intramuscularly (IM) as 3.75, 7.5, or 15 micrograms per dose; and inactivated influenza H1N1 vaccine without adjuvant, delivered intramuscularly as 7.5 or 15 micrograms per dose. All doses of the vaccine with or without adjuvant will be administered as a single 0.5 mL IM injection in the deltoid muscle of the preferred arm.

SUMMARY:
The purpose of this study is to see how the body reacts to different strengths of the H1N1 flu shot when it is given with or without an "adjuvant." An adjuvant is a substance that may cause the body to produce more antibodies when it is given with a vaccine. This study will also compare how age affects the body's response to the H1N1 flu shot. In this study, 3 strengths of the H1N1 flu shot will be tested combined with an adjuvant. In addition, 2 strengths of the H1N1 flu shot will be tested without adjuvant. Two H1N1 flu shots of the same strength, with or without adjuvant, will be given about 3 weeks apart. Participants will include up to 800 healthy adults, approximately 500 individuals ages 18-64 and 250 individuals greater than or equal to age 65. Study procedures include: physical exam, blood samples, completing a memory aid to record vaccine side effects, medications and daily oral temperature. Participants will be involved in study related procedures for up to 13 months.

DETAILED DESCRIPTION:
Recently, a novel swine-origin influenza A/H1N1 virus was identified as a significant cause of febrile respiratory illnesses in Mexico and the United States. It rapidly spread to many countries around the world, prompting the World Health Organization to declare a pandemic on June 11, 2009. Data from several cohorts in different age groups that received licensed trivalent seasonal influenza vaccines suggest that these vaccines are unlikely to provide protection against the new virus. Adults are more likely to have measurable levels of serum hemagglutination inhibition assay (HAI) or neutralizing antibody than are children. These data indicate the need to develop vaccines against the new H1N1 strain and suggest that different vaccine strategies (e.g., number of doses, need for adjuvant) may be appropriate for persons in different age groups. This protocol will explore antibody responses following vaccination with an inactivated influenza H1N1 virus vaccine at 3 different dose levels combined with AS03 adjuvant and at 2 different dose levels administered without adjuvant. This study will assess the immune response following a single dose of vaccine with or without AS03 adjuvant, to assess whether individuals have any pre-existing 'prime' immunity, such that the initial H1N1 vaccination serves as a boost, thus conferring a more rapid time to protection with the need for fewer doses. Antibody responses will be assessed at 8 days after each dose to evaluate the development of an anamnestic response. In addition, antibody responses will be assessed 21 days after each dose. The primary objectives are: safety, to assess the safety of inactivated H1N1 vaccine when administered at the 3.75 micrograms (mcg), 7.5 mcg, or 15 mcg dose combined with AS03 adjuvant and at the 7.5 mcg or 15 mcg dose administered without adjuvant; and immunogenicity, to assess the antibody response at Day 21 following a single dose of inactivated H1N1 vaccine when administered at 3.75 mcg, 7.5 mcg, or 15 mcg dose combined with AS03 adjuvant and at the 7.5 mcg or 15 mcg dose administered without adjuvant, stratified by age of recipient. The secondary objective is immunogenicity, to assess the antibody response following 2 doses of inactivated H1N1 vaccine when administered at the 3.75 mcg, 7.5 mcg, or 15 mcg dose combined with AS03 adjuvant and at the 7.5 mcg or 15 mcg dose administered without adjuvant, stratified by age of recipient. Participants will include up to 800 healthy adults who have no history of novel influenza H1N1 2009 infection or novel influenza H1N1 2009 vaccination. This is a randomized, double-blinded, Phase II study. Subjects will be randomized into 5 groups, stratified by age (150 subjects per dose group with 100 subjects in the 18-64 years of age stratum and 50 subjects in the greater than or equal to 65 years of age stratum), to receive intramuscular inactivated influenza H1N1 vaccine at 3.75 mcg, 7.5 mcg, or 15 mcg combined with AS03 adjuvant (Groups 1, 2, and 3, respectively) or at 7.5 mcg or 15 mcg without adjuvant (Groups 4 and 5, respectively). The vaccine, with and without adjuvant, will be administered at Day 0 and Day 21. Following immunization, safety will be measured by assessment of adverse events (AEs) through 21 days following the last vaccination (Day 42 for those receiving both doses and Day 21 for those who do not receive the second dose), serious adverse events (SAEs) and new-onset chronic medical conditions through 12 months post final vaccination (Day 365 after second vaccination), and reactogenicity to vaccine for 8 days (Day 0-7) following each vaccination. Immunogenicity testing will include HAI and neutralizing antibody.

ELIGIBILITY:
Inclusion Criteria:

1. Are males or non-pregnant females age 18 and older, inclusive.
2. Women of child-bearing potential (not surgically sterile via tubal ligation, bilateral oophorectomy or hysterectomy or who are not postmenopausal for greater than or equal to 1 year) must agree to practice adequate contraception that may include, but is not limited to, abstinence, monogamous relationship with vasectomized partner, barrier methods such as condoms, diaphragms, spermicides, intrauterine devices, and licensed hormonal methods during the study for at least 30 days following the last vaccination.
3. Are in good health, as determined by vital signs, medical history to ensure any existing medical diagnoses or conditions are stable and not considered clinically significant, and limited physical examination. A stable chronic medical condition is defined as no change in prescription medication, dose, or frequency of medication in the last 3 months and health outcomes of the specific disease are considered to be within acceptable limits in the last 6 months. Any change that is due to change of health care provider, insurance company etc, or that is done for financial reasons, as long as in the same class of medication will not be considered a violation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome will not be considered a violation of this inclusion criterion.
4. Have alanine aminotransferase (ALT) within normal range per local or site laboratory reference ranges.
5. Are able to understand and comply with planned study procedures.
6. Provide written informed consent prior to initiation of any study procedures.

Exclusion Criteria:

1. Have a known allergy to eggs or other components of the vaccine (including squalene based adjuvants, gelatin, formaldehyde, octoxinol, thimerosal, and chicken protein).
2. Have a positive urine or serum pregnancy test within 24 hours prior to vaccination (if female of childbearing potential), or women who are breastfeeding.
3. Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy (cytotoxic) within the preceding 36 months.
4. Have an active neoplastic disease or a history of any hematologic malignancy.
5. Have long term use of glucocorticoids including oral, parenteral or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months. (Nasal and topical steroids are allowed.)
6. Have a diagnosis of schizophrenia, bipolar disease, or other major psychiatric diagnosis.
7. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others, within the past 10 years.
8. Are receiving psychiatric drugs (aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, chlorprothixene, chlorpromazine, perphenazine, trifluopromazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate). Subjects who are receiving a single antidepressant drug and are stable for at least 3 months prior to enrollment, without de-compensating symptoms will be allowed to be enrolled in the study.
9. Have a history of receiving immunoglobulin or other blood product within the 3 months prior to vaccination in this study.
10. Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to vaccination in this study or expect to receive an experimental agent during this study (prior to the Day 386 clinic visit - 365 days after the second vaccination).
11. Have received any live licensed vaccines within 4 weeks or inactivated licensed vaccines within 2 weeks prior to vaccination in this study or plan receipt of such vaccines within 21 days following the second vaccination. This is inclusive of seasonal influenza vaccines.
12. Have an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe, or would interfere with the evaluation of responses.
13. Have a history of severe reactions following previous immunization with influenza virus vaccines.
14. Have an acute illness, including an oral temperature greater than 100.4 degrees Fahrenheit, within 3 days prior to vaccination.
15. Have any condition that would, in the opinion of the site investigator, place them at an unacceptable risk of injury or render them unable to meet the requirements of the protocol.
16. Participated in a novel influenza H1N1 2009 vaccine study in the past 2 years or have a history of novel influenza H1N1 2009 infection prior to enrollment.
17. Have known active human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C infection or autoimmune hepatitis.
18. Have a history of alcohol or drug abuse in the last 5 years.
19. Plan to travel outside of North America in the time between the first vaccination and 42 days following the first vaccination.
20. Have a history of Guillain-Barré Syndrome.
21. Have any condition that the investigator believes may interfere with successful completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 789 (Actual)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Stanford University - Stanford Hospital and Clinics - Pediatrics - Infectious Diseases, Stanford, California
  - Emory Vaccine Center - The Hope Clinic, Decatur, Georgia
  - University of Iowa - Vaccine Research & Education Unit, Iowa City, Iowa
  - University of Maryland School of Medicine - Center for Vaccine Development - Baltimore, Baltimore, Maryland
  - Cincinnati Children's Hospital Medical Center - Infectious Diseases, Cincinnati, Ohio
  - Group Health Research Institute - Seattle, Seattle, Washington
  - The University of Washington - Virology Research Clinic, Seattle, Washington

REFERENCES:
- [Result] Jackson LA, Chen WH, Stapleton JT, Dekker CL, Wald A, Brady RC, Edupuganti S, Winokur P, Mulligan MJ, Keyserling HL, Kotloff KL, Rouphael N, Noah DL, Hill H, Wolff MC. Immunogenicity and safety of varying dosages of a monovalent 2009 H1N1 influenza vaccine given with and without AS03 adjuvant system in healthy adults and older persons. J Infect Dis. 2012 Sep 15;206(6):811-20. doi: 10.1093/infdis/jis427. Epub 2012 Jul 10. PMID 22782949

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy adults age 18 and older recruited from existing volunteer populations and from the communities at large around the clinical sites. Participants were enrolled between 24Sep2009 and 16Nov2009.
Groups:
- 3.75 mcg H1N1 Vaccine + AS03 Adjuvant: Participants received 3.75 mcg H1N1 vaccine plus AS03 adjuvant on Day 0 and Day 21.
- 7.5 mcg H1N1 Vaccine + AS03 Adjuvant: Participants received 7.5 mcg H1N1 vaccine plus AS03 adjuvant on Day 0 and Day 21.
- 7.5 mcg H1N1 Vaccine Unadjuvanted: Participants received 7.5 mcg H1N1 vaccine unadjuvanted on Day 0 and Day 21.
- 15 mcg H1N1 Vaccine + AS03 Adjuvant: Participants received 15 mcg H1N1 vaccine plus AS03 adjuvant on Day 0 and Day 21.
- 15 mcg H1N1 Vaccine Unadjuvanted: Participants received 15 mcg H1N1 vaccine unadjuvanted on Day 0 and Day 21.
Period: Overall Study
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Started | 156 | 163 | 160 | 157 | 153
Completed | 151 | 159 | 155 | 150 | 151
Not Completed | 5 | 4 | 5 | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted | Total
Number analyzed (Participants) | 156 | 163 | 160 | 157 | 153 | 789
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 107 | 111 | 110 | 109 | 107 | 544
  >=65 years | 49 | 52 | 50 | 48 | 46 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (17.6) | 51.7 (18.0) | 51.6 (17.8) | 50.1 (18.3) | 52.1 (18.6) | 51.4 (18.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 84 | 93 | 85 | 72 | 423
  Male | 67 | 79 | 67 | 72 | 81 | 366
Region of Enrollment [Number; unit: participants]
  United States | 156 | 163 | 160 | 157 | 153 | 789

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Age 18 to 64 Years With 4-fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 8 Days Following the First Dose of H1N1 Vaccine
Description: Blood was collected from participants for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 8 post first H1N1 vaccination titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 8 titer was an increase by 4-fold or more.
Time Frame: Day 0 prior to vaccination and 8 days after the first H1N1 vaccination
Population: Participants who received the H1N1 vaccination and from whom blood was collected are included. One participant was excluded due to an eligibility deviation. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 106 | 110 | 110 | 107 | 107
Participants | 84 | 95 | 62 | 94 | 80

2. Primary Outcome: Number of Participants Age 18 to 64 Years With 4-fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 21 Days Following the First Dose of H1N1 Vaccine
Description: Blood was collected from participants for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 21 post first H1N1 vaccination titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 21 titer was an increase by 4-fold or more.
Time Frame: Day 0 prior to vaccination and 21 days after the first H1N1 vaccination
Population: Participants who received the H1N1 vaccination and from whom blood was collected within 7 days of the window are included. One participant was excluded due to eligibility deviation and two due to receipt of off-study vaccines. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 105 | 109 | 105 | 104 | 105
Participants | 90 | 96 | 72 | 96 | 86

3. Primary Outcome: Number of Participants Age 65 Years and Older With 4-fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 8 Days Following the First Dose of H1N1 Vaccine
Description: as for outcome 1
Time Frame: Day 0 prior to vaccination and 8 days after the first H1N1 vaccination
Population: Participants who received the H1N1 vaccination and from whom blood was collected are included. One participant was excluded due to influenza-like illness. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 49 | 52 | 50 | 47 | 46
Participants | 24 | 30 | 17 | 34 | 21

4. Primary Outcome: Number of Participants Age 65 Years and Older With 4-fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 21 Days Following the First Dose of H1N1 Vaccine
Description: as for outcome 2
Time Frame: Day 0 prior to vaccination and 21 days after the first H1N1 vaccination
Population: Participants who received the H1N1 vaccination and from whom blood was collected within 7 days of the window are included. One participant was excluded due to influenza-like illness. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 48 | 52 | 48 | 45 | 44
Participants | 32 | 37 | 19 | 37 | 24

5. Primary Outcome: Number of Participants Reporting Vaccine-associated Serious Adverse Events (SAEs)
Description: Serious adverse events included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required in-patient hospitalization or prolongation thereof; resulted in a congenital anomaly/birth defect; may have jeopardized the participant or required intervention to prevent one of these outcomes; or was described as Guillain-Barré Syndrome. Association to vaccination was determined by a study clinician licensed to make medical diagnoses.
Time Frame: Day 0 through Day 365 after the last vaccination
Population: All participants receiving the first vaccination are included in the safety cohort. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 156 | 163 | 160 | 157 | 153
Participants | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants Age 18 to 64 Years With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 8 Days Following the Second Dose of H1N1 Vaccine
Description: Blood was collected from all participants 8 days after second vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 8 after the second vaccination
Population: Participants who received both H1N1 vaccinations and from whom blood was collected are included. One participant was excluded due to eligibility deviation, one due to receipt of the wrong second dose, and two due to receipt of off-study vaccines. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 101 | 103 | 101 | 99 | 99
Participants | 98 | 100 | 83 | 96 | 82

7. Secondary Outcome: Number of Participants Age 18 to 64 Years With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 21 Days Following the Second Dose of H1N1 Vaccine
Description: Blood was collected from all participants 21 days after second vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 21 after the second vaccination
Population: Participants who received both H1N1 vaccinations and from whom blood was collected within 7 days of window are included. One participant was excluded due to eligibility deviation, one due to receipt of the wrong second dose, and two due to receipt of off-study vaccines. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 100 | 103 | 101 | 99 | 96
Participants | 98 | 100 | 80 | 97 | 79

8. Primary Outcome: Number of Participants With Hematology Laboratory Adverse Events After the First Vaccination
Description: Blood was drawn 8-10 days after vaccination to assess laboratory parameters at a central laboratory. Adverse events (AE) were any values that were Grade 1 or greater for the following parameters: prothrombin time (AE >12.6 seconds), partial thromboplastin time (>40.7 seconds), platelets (>=401,000 or <=129,000 cells/square millimeter), white blood cells (>10,800 or <3800 cells/microliter), neutrophils (>8000 or <1800 cells/microliter), and lymphocytes(>4100 or <850 cells/microliter). These parameters were not evaluated prior to enrollment as an assessment of eligibility.
Time Frame: 8-10 days after first vaccination
Population: Participants who received the first vaccination and had blood collected with results reported at the timepoint are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 151 | 159 | 159 | 151 | 149
Participants
  Prothrombin time | 2 | 1 | 0 | 1 | 1
  Partial thromboplastin time | 3 | 1 | 1 | 1 | 1
  Platelets | 1 | 3 | 2 | 2 | 6
  White blood cells | 3 | 6 | 8 | 7 | 12
  Neutrophils | 2 | 3 | 5 | 3 | 8
  Lymphocytes | 3 | 1 | 5 | 2 | 1

9. Primary Outcome: Number of Participants With Hematology Laboratory Adverse Events After the Second Vaccination
Description: as for outcome 8
Time Frame: 8-10 days after second vaccination
Population: Participants who received at least the first vaccination and had blood collection at the timepoint are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 150 | 158 | 155 | 155 | 147
Participants
  Prothrombin time | 1 | 2 | 0 | 1 | 1
  Partial thromboplastin time | 4 | 3 | 0 | 3 | 3
  Platelets | 3 | 2 | 2 | 3 | 2
  White blood cells | 8 | 5 | 9 | 8 | 9
  Neutrophils | 8 | 5 | 2 | 5 | 7
  Lymphocytes | 4 | 0 | 3 | 1 | 4

10. Primary Outcome: Number of Participants With Chemistry Laboratory Adverse Events After the First Vaccination
Description: Blood was drawn 8-10 days after vaccination to assess laboratory parameters at a central laboratory. Adverse events (AE) were any values that were Grade 1 or greater for the following parameters: sodium (AE >146 or <135 mEq/L), potassium (>5.3 or <3.5 mEq/L), creatinine (>1.4 mg/dL), Alanine transaminase (>52.7 U/L), Albumin (<3.2 g/dL), and total protein (<6.0 g/dL participants age 18-64 years, <5.8 g/dL participants age 65 years and older). These parameters were not evaluated prior to enrollment as an assessment of eligibility.
Time Frame: 8-10 days after first vaccination
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 155 | 161 | 160 | 156 | 153
Participants
  Sodium | 0 | 1 | 1 | 2 | 3
  Potassium | 2 | 1 | 2 | 1 | 1
  Creatinine | 5 | 6 | 4 | 2 | 3
  Alanine transaminase | 0 | 1 | 3 | 1 | 2
  Albumin | 0 | 0 | 0 | 0 | 0
  Total protein | 2 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants Age 18 to 64 Years With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 180 Days Following the Second Dose of H1N1 Vaccine
Description: Blood was collected from all participants 180 days after second vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 180 after the second vaccination
Population: Participants who received both H1N1 vaccinations and from whom blood was collected within 14 days of window are included. Two participants were excluded due to eligibility deviations, one due to receipt of the wrong second dose, and two due to receipt of off-study vaccines. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 98 | 103 | 99 | 96 | 97
Participants | 90 | 87 | 66 | 83 | 69

12. Secondary Outcome: Number of Participants Age 18 to 64 Years With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 270 Days Following the Second Dose of H1N1 Vaccine
Description: Blood was collected from all participants 270 days after second vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 270 after the second vaccination
Population: as for outcome 11
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 90 | 100 | 98 | 92 | 96
Participants | 71 | 71 | 58 | 71 | 62

13. Secondary Outcome: Number of Participants Age 65 Years and Older With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 8 Days Following the Second Dose of H1N1 Vaccine
Description: as for outcome 6
Time Frame: Day 8 after the second vaccination
Population: Participants who received both H1N1 vaccinations and from whom blood was collected are included. One participant was excluded due to influenza-like illness and one due to receipt of off-study vaccine. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 44 | 47 | 46 | 41 | 37
Participants | 37 | 43 | 29 | 39 | 23

14. Secondary Outcome: Number of Participants Age 65 Years and Older With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 21 Days Following the Second Dose of H1N1 Vaccine
Description: as for outcome 7
Time Frame: Day 21 after the second vaccination
Population: Participants who received both H1N1 vaccinations and from whom blood was collected within 7 days of window are included. One participant was excluded due to influenza-like illness and two due to receipt of off-study vaccines. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 44 | 47 | 46 | 40 | 37
Participants | 36 | 44 | 29 | 38 | 25

15. Secondary Outcome: Number of Participants Age 65 Years and Older With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 180 Days Following the Second Dose of H1N1 Vaccine
Description: as for outcome 11
Time Frame: Day 180 after the second vaccination
Population: Participants who received both H1N1 vaccinations and from whom blood was collected within 14 days of window are included. One participant was excluded due to influenza-like illness and two due to receipt of off-study vaccines. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 44 | 47 | 46 | 40 | 36
Participants | 29 | 36 | 26 | 36 | 18

16. Secondary Outcome: Number of Participants Age 65 Years and Older With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 270 Days Following the Second Dose of H1N1 Vaccine
Description: as for outcome 12
Time Frame: Day 270 after the second vaccination
Population: as for outcome 15
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 43 | 47 | 42 | 40 | 36
Participants | 21 | 30 | 16 | 30 | 13

17. Secondary Outcome: Number of Participants Age 18 to 64 Years With 4-fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 8 Days Following the Second Dose of H1N1 Vaccine
Description: Blood was collected from participants for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 8 post second H1N1 vaccination titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 8 titer was an increase by 4-fold or more.
Time Frame: Day 0 prior to vaccination and 8 days after the second H1N1 vaccination
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 101 | 103 | 101 | 99 | 99
Participants | 95 | 98 | 79 | 93 | 80

18. Primary Outcome: Number of Participants With Chemistry Laboratory Adverse Events After the Second Vaccination
Description: as for outcome 10
Time Frame: 8-10 days after second vaccination
Population: Participants who received at least the first vaccination and had blood collected with results reported at the timepoint are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 150 | 158 | 154 | 153 | 147
Participants
  Sodium | 1 | 0 | 2 | 2 | 0
  Potassium | 0 | 1 | 1 | 0 | 0
  Creatinine | 2 | 3 | 3 | 0 | 3
  Alanine transaminase | 1 | 1 | 1 | 2 | 0
  Albumin | 0 | 0 | 0 | 0 | 0
  Total protein | 1 | 0 | 0 | 0 | 1

19. Primary Outcome: Number of Participants Reporting Solicited Subjective Systemic Reactions After the First Vaccination
Description: Participants maintained a memory aid to record daily the occurrence of systemic symptoms of feverishness, malaise, myalgia, headache, nausea, chills, arthralgia, and shivering for 8 days (Day 0-7) after vaccination based on their interference with daily activities. Participants are counted if they reported experiencing the symptom at any severity on any of the 8 days.
Time Frame: Within 8 days (Day 0-7) post first vaccination
Population: Participants who received the first vaccination are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 156 | 163 | 160 | 157 | 153
Participants
  Feverishness | 15 | 18 | 5 | 22 | 10
  Malaise | 42 | 41 | 29 | 44 | 32
  Myalgia | 32 | 43 | 13 | 45 | 24
  Headache | 40 | 38 | 35 | 35 | 38
  Nausea | 12 | 9 | 7 | 12 | 10
  Chills | 17 | 15 | 5 | 12 | 12
  Arthralgia | 13 | 11 | 4 | 18 | 9
  Shivering | 7 | 9 | 3 | 7 | 5

20. Primary Outcome: Number of Participants Reporting Solicited Subjective Systemic Reactions After the Second Vaccination
Description: as for outcome 19
Time Frame: Within 8 days (Day 0-7) post second vaccination
Population: Participants who received the second vaccination are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 147 | 151 | 151 | 147 | 140
Participants
  Feverishness | 27 | 25 | 6 | 32 | 8
  Malaise | 47 | 41 | 17 | 40 | 19
  Myalgia | 38 | 39 | 10 | 35 | 14
  Headache | 35 | 47 | 27 | 31 | 21
  Nausea | 16 | 10 | 5 | 10 | 5
  Chills | 19 | 18 | 3 | 20 | 5
  Arthralgia | 11 | 17 | 6 | 13 | 9
  Shivering | 14 | 10 | 3 | 16 | 2

21. Secondary Outcome: Number of Participants Age 18 to 64 Years With 4-fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 21 Days Following the Second Dose of H1N1 Vaccine
Description: Blood was collected from participants for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 21 post second H1N1 vaccination titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 21 titer was an increase by 4-fold or more.
Time Frame: Day 0 prior to vaccination and 21 days after the second H1N1 vaccination
Population: Participants who received both H1N1 vaccinations and from whom blood was collected within 7 days of the window are included. One participant was excluded due to eligibility deviation, one due to receipt of the wrong second dose, and two due to receipt of off-study vaccines. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 100 | 103 | 101 | 99 | 96
Participants | 95 | 99 | 76 | 95 | 78

22. Secondary Outcome: Number of Participants Age 18 to 64 Years With 4-fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 180 Days Following the Second Dose of H1N1 Vaccine
Description: Blood was collected from participants for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 180 post second H1N1 vaccination titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 180 titer was an increase by 4-fold or more.
Time Frame: Day 0 prior to vaccination and 180 days after the second H1N1 vaccination
Population: Participants who received both H1N1 vaccinations and from whom blood was collected within 14 days of the window are included. Two participants were excluded due to eligibility deviations, one due to receipt of the wrong second dose, and two due to receipt of off-study vaccines. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 98 | 103 | 99 | 96 | 97
Participants | 82 | 83 | 56 | 79 | 65

23. Secondary Outcome: Number of Participants Age 18 to 64 Years With 4-fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 270 Days Following the Second Dose of H1N1 Vaccine
Description: Blood was collected from participants for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 270 post second H1N1 vaccination titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 270 titer was an increase by 4-fold or more.
Time Frame: Day 0 prior to vaccination and 270 days after the second H1N1 vaccination
Population: as for outcome 22
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 90 | 100 | 98 | 92 | 96
Participants | 65 | 69 | 49 | 66 | 55

24. Secondary Outcome: Number of Participants Age 65 Years and Older With 4-fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 8 Days Following the Second Dose of H1N1 Vaccine
Description: as for outcome 17
Time Frame: Day 0 prior to vaccination and 8 days after the second H1N1 vaccination
Population: as for outcome 13
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 44 | 47 | 46 | 41 | 37
Participants | 34 | 39 | 23 | 35 | 21

25. Secondary Outcome: Number of Participants Age 65 Years and Older With 4-fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 21 Days Following the Second Dose of H1N1 Vaccine
Description: as for outcome 21
Time Frame: Day 0 prior to vaccination and 21 days after the second H1N1 vaccination
Population: Participants who received both H1N1 vaccinations and from whom blood was collected within 7 days of the window are included. One participant was excluded due to influenza-like illness and two due to receipt of off-study vaccines. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 44 | 47 | 46 | 40 | 37
Participants | 33 | 41 | 23 | 36 | 23

26. Secondary Outcome: Number of Participants Age 65 Years and Older With 4-fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 180 Days Following the Second Dose of H1N1 Vaccine
Description: as for outcome 22
Time Frame: Day 0 prior to vaccination and 180 days after the second H1N1 vaccination
Population: Participants who received both H1N1 vaccinations and from whom blood was collected within 14 days of the window are included. One participant was excluded due to influenza-like illness and two due to receipt of off-study vaccines. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 44 | 47 | 46 | 40 | 36
Participants | 25 | 31 | 21 | 29 | 15

27. Secondary Outcome: Number of Participants Age 65 Years and Older With 4-fold or Greater Hemagglutination Inhibition Assay (HAI) Antibody Titer Increases Against the Influenza H1N1 2009 Virus 270 Days Following the Second Dose of H1N1 Vaccine
Description: as for outcome 23
Time Frame: Day 0 prior to vaccination and 270 days after the second H1N1 vaccination
Population: as for outcome 26
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 43 | 47 | 42 | 40 | 36
Participants | 19 | 23 | 12 | 22 | 11

28. Primary Outcome: Number of Participants Reporting Fever After the First Vaccination
Description: Participants were provided a thermometer and a memory aid to record daily oral temperatures for 8 days (Day 0-7) after vaccination. Participants are counted as experiencing fever if they reported oral temperatures of 38 degrees Celsius or higher on any of the 8 days.
Time Frame: Within 8 days (Day 0-7) post first vaccination
Population: Participants who received the first vaccination and reported oral temperatures during the time period are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 156 | 163 | 159 | 156 | 153
Participants | 2 | 4 | 0 | 3 | 0

29. Primary Outcome: Number of Participants Reporting Fever After the Second Vaccination
Description: as for outcome 28
Time Frame: Within 8 days (Day 0-7) post second vaccination
Population: Participants who received the second vaccination and reported oral temperatures during the time period are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 147 | 151 | 151 | 147 | 140
Participants | 8 | 4 | 0 | 6 | 0

30. Primary Outcome: Number of Participants Reporting Solicited Subjective Local Reactions After the First Vaccination
Description: Participants maintained a memory aid to record daily the occurrence of local symptoms of pain, tenderness and swelling for 8 days (Day 0-7) after vaccination based on their interference with daily activities. Participants are counted if they reported experiencing the symptom at any severity on any of the 8 days.
Time Frame: Within 8 days (Day 0-7) post first vaccination
Population: Participants who received the first vaccination are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 156 | 163 | 160 | 157 | 153
Participants
  Pain | 90 | 96 | 25 | 90 | 35
  Tenderness | 122 | 130 | 37 | 115 | 55
  Swelling | 33 | 28 | 20 | 31 | 27

31. Primary Outcome: Number of Participants Reporting Solicited Subjective Local Reactions After the Second Vaccination
Description: as for outcome 30
Time Frame: Within 8 days (Day 0-7) post second vaccination
Population: Participants who received the second vaccination are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 147 | 151 | 151 | 147 | 140
Participants
  Pain | 73 | 82 | 16 | 66 | 28
  Tenderness | 104 | 112 | 37 | 100 | 51
  Swelling | 26 | 19 | 24 | 27 | 20

32. Primary Outcome: Number of Participants Reporting Solicited Quantitative Local Reactions After the First Vaccination
Description: Participants maintained a memory aid to record daily the occurrence of local reactions of redness and swelling for 8 days (Day 0-7) after vaccination. If the reaction was present, the maximum diameter was measured in millimeters (mm). Participants are counted if they were reported as experiencing the reaction with any measurement greater than 0 mm on any of the 8 days.
Time Frame: Within 8 days (Day 0-7) post first vaccination
Population: Participants who received the first vaccination are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 156 | 163 | 160 | 157 | 153
Participants
  Redness | 41 | 36 | 33 | 44 | 40
  Swelling | 36 | 30 | 22 | 32 | 28

33. Primary Outcome: Number of Participants Reporting Solicited Quantitative Local Reactions After the Second Vaccination
Description: as for outcome 32
Time Frame: Within 8 days (Day 0-7) post second vaccination
Population: Participants who received the second vaccination are included. Analyses are as treated.
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 147 | 151 | 151 | 147 | 140
Participants
  Redness | 28 | 29 | 30 | 40 | 30
  Swelling | 27 | 17 | 25 | 30 | 23

34. Primary Outcome: Number of Participants Age 18 to 64 Years With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 8 Days Following the First Dose of H1N1 Vaccine
Description: Blood was collected from all participants 8 days after vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 8 after the first vaccination
Population: Participants who received the H1N1 vaccination and from whom blood was collected at the timepoint are included. One participant was excluded due to eligibility deviation. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 106 | 110 | 110 | 107 | 107
Participants | 91 | 96 | 67 | 98 | 82

35. Primary Outcome: Number of Participants Age 18 to 64 Years With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 21 Days Following the First Dose of H1N1 Vaccine
Description: Blood was collected from all participants 21 days after vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 21 after the first vaccination
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 105 | 109 | 105 | 104 | 105
Participants | 95 | 97 | 78 | 99 | 87

36. Primary Outcome: Number of Participants Age 65 Years and Older With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 8 Days Following the First Dose of H1N1 Vaccine
Description: as for outcome 34
Time Frame: Day 8 after the first vaccination
Population: Participants who received the H1N1 vaccination and from whom blood was collected at the timepoint are included. One participant was excluded due to influenza-like illness. Analyses are as treated. This outcome restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 49 | 52 | 50 | 47 | 46
Participants | 26 | 36 | 25 | 38 | 25

37. Primary Outcome: Number of Participants Age 65 Years and Older With a Serum Hemagglutination Inhibition Assay (HAI) Antibody Titer of 1:40 or Greater Against the H1N1 2009 Virus 21 Days Following the First Dose of H1N1 Vaccine
Description: as for outcome 35
Time Frame: Day 21 after the first vaccination
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Number analyzed (Participants) | 48 | 52 | 48 | 45 | 44
Participants | 34 | 42 | 27 | 40 | 27

ADVERSE EVENTS:
Time Frame: Solicited events were collected for 8 days after each vaccination, unsolicited events through 21 days after last vaccination, and serious adverse events and new onset chronic medical conditions through 365 days after last vaccination.
Description: For events solicited on a Memory Aid in the 8 days after vaccination, a participant was considered to have one event if it was reported as experienced at any time in the 8 day period.
Arm/Group | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant | 7.5 mcg H1N1 Vaccine Unadjuvanted | 15 mcg H1N1 Vaccine + AS03 Adjuvant | 15 mcg H1N1 Vaccine Unadjuvanted
Serious Adverse Events (participants affected / at risk) | 6/156 | 7/163 | 12/160 | 8/157 | 8/153
Other Adverse Events (participants affected / at risk) | 147/156 | 157/163 | 124/160 | 146/157 | 130/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant (N=156) | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant (N=163) | 7.5 mcg H1N1 Vaccine Unadjuvanted (N=160) | 15 mcg H1N1 Vaccine + AS03 Adjuvant (N=157) | 15 mcg H1N1 Vaccine Unadjuvanted (N=153)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric bypass (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aqueductal stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cervical myelopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder prolapse (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal laminectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial septal defect repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dementia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Implantable defibrillator insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemophilus sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 3.75 mcg H1N1 Vaccine + AS03 Adjuvant (N=156) | 7.5 mcg H1N1 Vaccine + AS03 Adjuvant (N=163) | 7.5 mcg H1N1 Vaccine Unadjuvanted (N=160) | 15 mcg H1N1 Vaccine + AS03 Adjuvant (N=157) | 15 mcg H1N1 Vaccine Unadjuvanted (N=153)
Blood pressure systolic increased (Investigations) | 2 (2) | 3 (3) | 3 (3) | 8 (8) | 5 (5)
Injection site haematoma (General disorders) | 10 (10) | 4 (4) | 9 (10) | 5 (5) | 8 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 8 (10) | 8 (8) | 3 (3) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 15 (18) | 17 (18) | 20 (22) | 16 (17) | 22 (25)
Pyrexia (General disorders) | 8 (10) | 7 (8) | 0 (0) | 9 (9) | 0 (0)
Feeling hot (General disorders) | 35 (42) | 35 (43) | 11 (11) | 44 (54) | 15 (18)
Malaise (General disorders) | 66 (89) | 67 (82) | 37 (46) | 61 (84) | 44 (51)
Myalgia (Musculoskeletal and connective tissue disorders) | 55 (70) | 67 (82) | 22 (23) | 60 (80) | 32 (38)
Headache (Nervous system disorders) | 59 (75) | 68 (85) | 54 (62) | 47 (66) | 46 (59)
Nausea (Gastrointestinal disorders) | 22 (28) | 19 (19) | 11 (12) | 19 (22) | 15 (15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 (24) | 27 (28) | 9 (10) | 26 (31) | 14 (18)
Chills (General disorders) | 29 (36) | 28 (33) | 7 (8) | 30 (32) | 17 (17) — Solicited as "chills"
Chills (General disorders) | 17 (21) | 19 (19) | 6 (6) | 22 (23) | 7 (7) — Solicited as "shivering"
Injection site pain (General disorders) | 101 (163) | 117 (178) | 33 (41) | 102 (156) | 47 (63)
Tenderness (General disorders) | 138 (226) | 141 (242) | 52 (74) | 128 (215) | 70 (106) — Tenderness was solicited as a reaction at the vaccination site.
Injection site erythema (General disorders) | 54 (69) | 52 (65) | 51 (63) | 63 (84) | 53 (70)
Injection site swelling (functional grading) (General disorders) | 46 (59) | 36 (47) | 33 (44) | 47 (58) | 37 (47) — Injection site swelling was solicited separately for functional grading of impact on daily activities and as a measured reaction.
Injection site swelling (measured) (General disorders) | 48 (63) | 40 (47) | 37 (47) | 51 (62) | 42 (51) — Injection site swelling was solicited separately for functional grading of impact on daily activities and as a measured reaction.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less